CLINICAL TRIAL: NCT04286204
Title: New Information and Communication Technologies (ICT´s) in Basic Life Support Training for Non-medical Students: Educational Trial.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: For COVID -19 pandemic, all participants (undergradueted students) can not completed the research protocol.
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SIIU 2019-28530
Record Dates: First submitted 2019-12-13; First posted 2020-02-26 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2021-04

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
Keywords: Cardiac Arrest; Basic Life Support; New Information and Communication Technologies
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic Life Support Training based on ICTs (Experimental): It will be conformed with students from one highschool random selected. They will receive a basic life support training based on Information and communication technologies.
  Interventions: Other: Basic Life Support training based on ICTs
- Classic Basic Life Support Training (Active Comparator): It will be conformed with students from another highschool random selected. They will receive a full and conventional basic life support training based on American and Hear Association recommendations.
  Interventions: Other: Classic Basic Life Support training

INTERVENTIONS:
Other: Basic Life Support training based on ICTs — This intervention is defined as a self-training course consisting of a 5-minute educational video in basic life support and a Kit with the elements to build the home dummy and the home DEA allowing integrally students to develop the steps as the video. The Kit will be delivered at the beginning of the study and every month the necessary materials will be complemented. The strategy will be carried out by the students every month and supervised by their teachers. Students will have constant access to an educational platform based on ICTs.
  Arms: Basic Life Support Training based on ICTs
Other: Classic Basic Life Support training — It is defined as a module carried out by trained personnel in basic resuscitation (pre-hospital care program staff of the UdeA medical school), which includes two subcomponents of the conventional BLS course that are basic resuscitation and DEA in adults. The duration of the subcomponents is a theoretical part of 30 minutes and a practical part in a low fidelity simulator with 1.5 hours duration.
  Arms: Classic Basic Life Support Training

SUMMARY:
With the increase in life expectancy of the general population and advances in medicine, there is now a population with a higher amount of cardiovascular diseases that lead to an increased risk of sudden cardiac arrest. In most cases, this occurs in extra-hospital settings such as family homes, shopping centres, public transport and before people without any knowledge or training in basic life support. On the other hand, for every minute that passes without adequate attention of the victim, the probability of surviving or continuing to live with neurological severe sequelae decreases by 10%.

In developed countries, public policies have been created to encourage basic life support education to the general population. In Colombia, because of the high prevalence of these diseases and the need for public health strategies, a law was issued to provide access to automatic external defibrillators (AEDs) in public places. However, it has not been developed strategies for education on this subject.

For that reason, the investigators created an educational strategy of self-learning, which consists of a complete basic life support course based in new Information and Communication technologies with tools to manufacture a mannequin and a homemade DEA, which will allow continuous training, with a very low cost compared to traditional life support training.

The clinical trial will compare that two educational strategies, evaluating as primary aid, which approach has higher knowledge retention of life support chain at 6 months in students after the workshop. As secondary objectives, the investigators would evaluate the efficient in terms of response times, costs and student satisfaction.

This study will be carried out in high school students from two different high schools, without prior training in Life support. Both strategies will be distributed randomly. The experimental group will carry out the self-learning strategy based on ICT (Information and Communication Technologies), with which they will be retrained every month, and the control group will carry out the conventional training only once as usual. Subsequently, each of the objectives will be evaluated at six months.

It is proposed that the self-learning strategy is superior compared to conventional training, requiring fewer resources to perform it and allows constant retraining, which improves retention and quality in a resuscitation process.

ELIGIBILITY:
Inclusion Criteria:

* Senior students over 14 years in high school.

Exclusion Criteria:

* Cognitive disorders.
* Cardiovascular o pulmonary diseases.
* Any condition that prevents physical activities.
* To have any previous training in basic life support.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality in survival chain in basic life support | 6 months
  It will be a composed outcome of 6 aspects in a check list and the student must comply ALL item to consider as a positive result in good quality in basic life support, the items are:
  I. Recognition of a person in cardiorespiratory arrest II. Activate the survival chain to survive III. Start chest compressions during or after activating the chain. IV. Chest compressions between 100-120 V. Proper use of AED VI. No interruptions should made during the thoracic compressions cycle. The result will be presented in proportion of students who completed ALL previous items.

SECONDARY OUTCOMES:
Time of survival chain activation | 6 months
  Time in seconds that takes the student to perform the following components of the survival chain:
  * Identification of the victim
  * Emergency system activation.
  * Start of chest compressions.
  * Implementation of the AED strategy.
Student Satisfaction | 6 months
  The satisfaction scale will be applied to all students. We will use a satisfaction scale developed and validated in Oviedo´s University, Asturias, Spain. It is a seven items scale. Each item is evaluated in 4 points Likert scale. The minimum value is 1, and the maximum value is 4 for each item.
  We will evaluate these scale independently and present results in number and percentage en each item.
Costs | 6 months
  We will evaluate the cost in US dolar of each intervention in the different activities related to executions of the interventions in each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Villa-Velasquez, Dr, Principal Investigator — Univeridad de Antioquia's Professor
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Result] Meissner TM, Kloppe C, Hanefeld C. Basic life support skills of high school students before and after cardiopulmonary resuscitation training: a longitudinal investigation. Scand J Trauma Resusc Emerg Med. 2012 Apr 14;20:31. doi: 10.1186/1757-7241-20-31. PMID 22502917
- [Result] Li Q, Zhou RH, Liu J, Lin J, Ma EL, Liang P, Shi TW, Fang LQ, Xiao H. Pre-training evaluation and feedback improved skills retention of basic life support in medical students. Resuscitation. 2013 Sep;84(9):1274-8. doi: 10.1016/j.resuscitation.2013.04.017. Epub 2013 May 9. PMID 23665155
- [Result] Blewer AL, Leary M, Esposito EC, Gonzalez M, Riegel B, Bobrow BJ, Abella BS. Continuous chest compression cardiopulmonary resuscitation training promotes rescuer self-confidence and increased secondary training: a hospital-based randomized controlled trial*. Crit Care Med. 2012 Mar;40(3):787-92. doi: 10.1097/CCM.0b013e318236f2ca. PMID 22080629
- [Result] Smith KK, Gilcreast D, Pierce K. Evaluation of staff's retention of ACLS and BLS skills. Resuscitation. 2008 Jul;78(1):59-65. doi: 10.1016/j.resuscitation.2008.02.007. Epub 2008 Apr 10. PMID 18406037
- [Result] de Ruijter PA, Biersteker HA, Biert J, van Goor H, Tan EC. Retention of first aid and basic life support skills in undergraduate medical students. Med Educ Online. 2014 Nov 6;19:24841. doi: 10.3402/meo.v19.24841. eCollection 2014. PMID 25382803
- [Result] Pande S, Pande S, Parate V, Pande S, Sukhsohale N. Evaluation of retention of knowledge and skills imparted to first-year medical students through basic life support training. Adv Physiol Educ. 2014 Mar;38(1):42-5. doi: 10.1152/advan.00102.2013. PMID 24585468
- [Result] Einspruch EL, Lynch B, Aufderheide TP, Nichol G, Becker L. Retention of CPR skills learned in a traditional AHA Heartsaver course versus 30-min video self-training: a controlled randomized study. Resuscitation. 2007 Sep;74(3):476-86. doi: 10.1016/j.resuscitation.2007.01.030. Epub 2007 Apr 17. PMID 17442479
- [Result] Girish M, Rawekar A, Jose S, Chaudhari U, Nanoti G. Utility of Low Fidelity Manikins for Learning High Quality Chest Compressions. Indian J Pediatr. 2018 Mar;85(3):184-188. doi: 10.1007/s12098-017-2473-3. Epub 2017 Nov 20. PMID 29152687
- [Result] Jones I, Whitfield R, Colquhoun M, Chamberlain D, Vetter N, Newcombe R. At what age can schoolchildren provide effective chest compressions? An observational study from the Heartstart UK schools training programme. BMJ. 2007 Jun 9;334(7605):1201. doi: 10.1136/bmj.39167.459028.DE. Epub 2007 Apr 27. PMID 17468118
- [Result] Boet S, Bould MD, Pigford AA, Rossler B, Nambyiah P, Li Q, Bunting A, Schebesta K. Retention of Basic Life Support in Laypeople: Mastery Learning vs. Time-based Education. Prehosp Emerg Care. 2017 May-Jun;21(3):362-377. doi: 10.1080/10903127.2016.1258096. Epub 2017 Jan 6. PMID 28059603
- [Result] Pedersen TH, Kasper N, Roman H, Egloff M, Marx D, Abegglen S, Greif R. Self-learning basic life support: A randomised controlled trial on learning conditions. Resuscitation. 2018 May;126:147-153. doi: 10.1016/j.resuscitation.2018.02.031. Epub 2018 Mar 6. PMID 29522830
- [Result] Kanstad BK, Nilsen SA, Fredriksen K. CPR knowledge and attitude to performing bystander CPR among secondary school students in Norway. Resuscitation. 2011 Aug;82(8):1053-9. doi: 10.1016/j.resuscitation.2011.03.033. Epub 2011 Apr 13. PMID 21531067